CLINICAL TRIAL: NCT00053781
Title: A Phase II Study Of Perifosine (D-21266) In Previously Untreated Patients With Metastatic Or Recurrent Malignant Melanoma
Brief Title: Perifosine in Treating Patients With Metastatic or Recurrent Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I156; CAN-NCIC-IND156 (Other: PDQ); CDR0000269475 (Other: PDQ)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: perifosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of perifosine in treating patients who have metastatic or recurrent malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of perifosine, in terms of response rate, in previously untreated patients with metastatic or recurrent malignant melanoma.
* Assess the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral perifosine daily on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) or partial response (PR) receive 2 additional courses after documentation of CR or stable PR (i.e., no further tumor shrinkage).

Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma
* Metastatic or recurrent disease deemed incurable by standard therapies
* Clinically and/or radiologically documented disease by at least 1 site that is unidimensionally measurable as follows:

  * At least 20 mm by x-ray or physical exam
  * At least 10 mm by spiral CT scan
  * At least 20 mm by non-spiral CT scan
  * Bone lesions are not considered measurable
  * Outside previously irradiated area unless evidence of progression or new lesions within irradiated field
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 2.5 times ULN

Renal

* Creatinine no greater than ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions to compounds of similar chemical or biological composition to perifosine
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No ongoing or active infection
* No other concurrent uncontrolled medical illness, psychiatric illness, or social situation that would preclude study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior adjuvant immunotherapy
* No prior immunotherapy for recurrent/metastatic disease

Chemotherapy

* No prior chemotherapy (including regional therapy)
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy (except for low-dose, nonmyelosuppressive radiotherapy)

Surgery

* At least 4 weeks since prior major surgery

Other

* No other concurrent anticancer therapy or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-06-20 (Actual); Primary Completion 2004-09-14 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald S. Ernst, MD, FRCPC, Study Chair — London Health Sciences Centre
Locations (6):
- Canada (6):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital at University Health Network, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ernst DS, Eisenhauer E, Wainman N, Davis M, Lohmann R, Baetz T, Belanger K, Smylie M. Phase II study of perifosine in previously untreated patients with metastatic melanoma. Invest New Drugs. 2005 Dec;23(6):569-75. doi: 10.1007/s10637-005-1157-4. PMID 16034524